CLINICAL TRIAL: NCT04275193
Title: The Safety and Efficacy of the Traditional Chinese Medicine Zishenqing in Subjects With Active Systemic Lupus Erythematosus
Brief Title: The Safety and Efficacy of Zishenqing in Subjects With Active Systemic Lupus Erythematosus
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai University of Traditional Chinese Medicine (Other)
Collaborators: RenJi Hospital (Other)
Responsible Party: Principal Investigator, maojianchun, Professor, Shanghai University of Traditional Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: Zishenqing
Record Dates: First submitted 2020-02-12; First posted 2020-02-19 (Actual); Last update posted 2020-04-28 (Actual); Status verified 2020-04

CONDITIONS: Systemic Lupus Erythematosus
Keywords: Safety; Efficacy; Systemic Lupus Erythematosus
MeSH Terms: conditions — Lupus Erythematosus, Systemic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Zishenqing (Experimental): The original treatment and Zishenqing 1Co by mouth,twice a day for 12 weeks
  Interventions: Drug: Zishenqing
- Placebo (Placebo Comparator): The original treatment and Zishenqing simulator 1Co by mouth,twice a day for 12 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Zishenqing — Zishenqing Granule
  Other Names: Zishenqingqi
  Arms: Zishenqing
Drug: Placebo — Granule manufactured to mimic Zishenqing(containing 10% composition)
  Other Names: Placebo(for Zishenqing)
  Arms: Placebo

SUMMARY:
This study evaluates the safety and efficacy of the traditional chinese medicine Zishenqing in the treatment of active systemic lupus erythematosus.

DETAILED DESCRIPTION:
This study will be a multicenter, randomized, double-blind, placebo parallel controlled clinical trial with a course of 12 weeks.

1. Multicenter: During the study period, it will be decided whether to increase the improvement progress of the research unit according to whether it will be difficult to join the group and the overall progress, so as to complete the clinical study on time in accordance with the research plan.
2. Random scheme: In this study, a dynamic random variance minimization random scheme will be adopted. Considering the two influencing factors of SLEDAI score and complement level, the DAS for Interactive Web Response System(IWRS) will be used to calculate and distribute random numbers and dispensing drugs.
3. Control drug: Placebo will be used as control in this trial.
4. Blind method: The Zishenqing simulator will be prepared by double-blind design, the dosage form, appearance, size, color and smell will be consistent with the experimental drug, and the test process will be in a double-blind state.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who qualify for the diagnosis of systemic lupus erythematosus according to the American college of rheumatology's 1997 revised classification criteria for systemic lupus erythematosus;
2. For inpatient or out-patient with good compliance, sign the informed consent before the test;
3. Sledai score during screening period≤10;
4. Maintain a stable standard treatment regimen for at least 30 days before the first day (that is, the date of administration of the intervention drug). Standard treatment regimens refer to the stable use of any of the following (alone or in combination): corticosteroids, hydroxychloroquine, non-steroidal anti-inflammatory drugs, other immunosuppressants or immunomodulators (including azathioprine, mycophenolate ester, cyclophosphamide, methotrexate, leflunomide, tacrolimus, cyclosporine);

Exclusion Criteria:

1. Severe lupus nephritis requiring hemodialysis or high-dose glucocorticoid treatment in the last 2 months;
2. Central nervous system diseases (including epilepsy, psychosis, organic encephalopathy syndrome, cerebrovascular accident, encephalitis, central nervous system vasculitis) caused by SLE or non-SLE in the last 2 months;
3. Patients with severe heart, liver and kidney diseases and disease history of important organs, blood and endocrine system;

   Evaluation criteria of severity:
   1. Alanine aminotransferase(ALT) and Aspartate aminotransferase(AST)≥3 times the upper limit of normal;
   2. Glomerular filtration rate(GFR)<30ml/min;
   3. White Blood Cell(WBC)<2.0×10^9/l;
   4. Platelet(PLT)<50×10^9/l;
4. Immunodeficiency, uncontrolled infection and active or recurrent peptic ulcer;
5. Pregnant and lactating women;
6. Anaphylaxis: allergic to traditional Chinese medicine;
7. The investigator considered it inappropriate to participate in this study;
8. Participate in other clinical trials during the screening period.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 118 (Estimated)
Dates: Start 2019-10-22 (Actual); Primary Completion 2022-03-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Lupus Quality of Life (LupusQoL) | 12weeks
  Self reported the quality of life in patients with systemic lupus erythematosus.LupusQoL is made up of five parts((physical health, pain, planning, emotional health, and fatigue) and has a total of 34 questions.Each question is scored0-4,yielding a total between 0 and 136.

SECONDARY OUTCOMES:
The 36-item shot form health survey(SF-36) | 12weeks
  As a concise health questionnaire, SF-36 comprehensively summarizes the quality of life of the subjects from eight aspects: physiological function, physiological function, physical pain, general health status, energy, social function, emotional function and mental health.
Systemic lupus erythematosus disease activity index(SLEDAI) | 12weeks
  SLEDAI scores are used to determine the activity of SLE.SLEDAI consists of 24 clinical and laboratory projects with different weights（0:no activity;1-5:mild activity;6-10:moderate activity;11-19:severe activity;≥20:extremely severe activity).

CONTACTS AND LOCATIONS:
Overall Officials: Liangjing Lv, Ph.D, Study Chair — RenJi Hospital; Huanru Qu, Ph.D, Study Chair — Longhua Hospital; Zhujing Zhu, Ph.D, Study Chair — Longhua Hospital; Ruru Guo, Ph.D, Study Chair — RenJi Hospital; Zhongping Xu, Master, Study Chair — Longhua Hospital
Locations (1):
- Longhua Hospital Affiliated to Shanghai University of Traditional Chinese Medicine, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No